CLINICAL TRIAL: NCT03651713
Title: Effect of Short-Term Glucose Loading on Vascular Function
Brief Title: Hyperglycemia, Exercise, and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Darren P Casey, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201807752
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Endothelial Function; Hyperglycemia
Keywords: exercise; glucose; vascular function
MeSH Terms: conditions — Hyperglycemia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLU+EX (Experimental): Subjects will consume a 75g glucose beverage three times daily for seven days while participating in five structured aerobic exercise sessions throughout the experimental protocol.
  Interventions: Behavioral: GLU+EX
- GLU (Active Comparator): Subjects will consume a 75g glucose beverage three times daily for seven days without participating in structured aerobic exercise.
  Interventions: Dietary Supplement: GLU

INTERVENTIONS:
Behavioral: GLU+EX — Subjects will complete 45 minutes of recumbent cycling at 60-65% of age-predicted maximal heart rate five times over seven days while ingesting a 75g glucose beverage three times daily.
  Arms: GLU+EX
Dietary Supplement: GLU — Subjects will consume a 75g glucose beverage three times daily over a seven-day period.
  Arms: GLU

SUMMARY:
The main purpose of this study is to determine if exercise preserves vascular function during hyperglycemia. All subjects will consume a sugary beverage three times daily for seven days. Subjects will be randomly assigned to either the glucose with (GLU+EX) or without (GLU) structured exercise group.

DETAILED DESCRIPTION:
Acute (oral glucose tolerance test) and chronic (type 2 diabetes) hyperglycemia are associated with impaired endothelial function. Both a single bout of exercise and chronic exercise training are associated with improvements in vascular endothelial function. It remains unknown if exercise can preserve vascular endothelial function during hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

- Healthy young men 18-35 years of age.

Exclusion Criteria:

* Hypertension,
* Hyperlipidemia,
* Smoking,
* Heart disease,
* Chest pain upon exertion,
* Previous heart surgeries or history of arrhythmias,
* Diabetes,
* Obesity (body mass index ≥30kg/m2),
* Kidney disease,
* Pulmonary disease,
* Autonomic disorders,
* Individuals whom engage in structured exercise (≥30min, ≥2d/wk),
* Current use of medications which influence outcome measures

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Vascular Endothelial Function | Before and after the seven-day intervention in both groups.
  Brachial artery flow-mediated dilation (%), measured via Doppler ultrasound, will be assessed before and after the intervention.

SECONDARY OUTCOMES:
Central Blood Pressure | Before and after the seven-day intervention in both groups.
  Aortic blood pressure will be derived from radial artery pressure wave measurements (via applanation tonometry) during resting conditions.

OTHER OUTCOMES:
Physical Activity | Continuously throughout the seven-day intervention.
  Steps per day will be recorded via accelerometry throughout the intervention in both groups.
Caloric Consumption | Continuously throughout the seven-day intervention.
  Subjects will record their dietary intake throughout the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Education Building, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No